CLINICAL TRIAL: NCT07163026
Title: Comparison of Analgesic Efficacy of Erector Spinae Plane Block and External Oblique-Intercostal Plane Block in Patients Undergoing Open Ventral Hernia Repair
Brief Title: Comparison of Two Plane Blocks Used in Open Ventral Hernia Repair Operations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Munire BABAYIGIT, Associate Professor, Ankara Ataturk Sanatorium Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SanatoryumEAH-AK-02
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Ventral Hernia; Postoperative Pain; Postoperative Nausea; Postoperative Vomiting
Keywords: erector spinae plane block; external oblique intercostal plane block; bupivacain
MeSH Terms: conditions — Hernia, Ventral; Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Block provider doesn't know peroperative process and the patient's postoperative assesment. Anesthesia provider doesn't know the block type and the patient's postoperative assesment. Outcomes assessor doesn't know about the block type and intraoperative process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESPB Group (Active Comparator): Erector spinae plane block will be applied to the patients in this group.
  Interventions: Procedure: Erector Spine Plane Block
- EOIPB Group (Sham Comparator): External Oblique - Intercostal Plane block will be applied to the patients in this group.
  Interventions: Procedure: External Oblique - Intercostal Plane Block

INTERVENTIONS:
Procedure: Erector Spine Plane Block — Bilateral erector spinae plane block was performed under aseptic conditions at the T7 vertebral level using ultrasound guidance with a convex probe. An 80-mm peripheral nerve block needle was inserted 3-4 cm lateral to the midline with an in-plane approach to the fascial plane deep to the erector spinae muscle. After negative aspiration and hydrodissection with 1-3 ml of saline, 30 ml of 0.25% bupivacaine was injected on each side, with craniocaudal spread confirmed by ultrasound. Patients were then positioned for surgery.
  Arms: ESPB Group
Procedure: External Oblique - Intercostal Plane Block — Bilateral external oblique-intercostal plane block was performed under aseptic conditions by identifying the 6th and 7th ribs along the midclavicular line. Using ultrasound guidance with the probe placed parallel to the midclavicular line, the ribs, intercostal muscles, external oblique muscle, and pleura were visualized. A 50-mm block needle was advanced craniocaudally into the plane between the external oblique and intercostal muscles. After negative aspiration and hydrodissection with 1-3 ml saline, 30 ml of 0.25% bupivacaine was injected on each side, with craniocaudal spread confirmed by ultrasound. Patients were then positioned for surgery.
  Arms: EOIPB Group

SUMMARY:
The aim of this study is to compare the postoperative analgesic efficacy of bilateral erector spinae plane block and bilateral external oblique-intercostal plane block in patients undergoing open ventral hernia repair.

DETAILED DESCRIPTION:
The effectiveness of trunk blocks applied at equivalent doses will be evaluated in order to most effectively treat postoperative pain, minimize nausea and vomiting, and optimize the comfort of patients during the postoperative period after open ventral hernia repair operations. The methods used in this study are proven safe in ventral hernia repair surgery and other abdominal surgeries, and are routinely performed in our clinic. The procedures performed pose no additional risks to patients compared to routine procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for open ventral hernia repair under general anesthesia
* Patients with ASA scores (American Society of Anesthesiologists) 1 and 2
* Patients with a body mass index between 18.5 and 34.9

Exclusion Criteria:

* Patients scheduled for open ventral hernia repair under spinal or epidural anesthesia
* Patients who have previously undergone spine surgery.
* Patients with known local anesthetic allergy
* Pregnant women
* Mentally uncooperative patients
* Patients with a history of chronic analgesic use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Tramadol Consumption | 24 hours
  The primary endpoint of the study was whether tramadol consumption in the first 24 hours was significantly different between groups.

SECONDARY OUTCOMES:
Remifentanil Consumption | 1 hour
  The amount of remifentanil consumption required to maintain normal vital signs during the intraoperative period.

OTHER OUTCOMES:
Pain Scores | 24 hours
  Difference between pain scores according to Visual Analog Scale at the 2nd and 24th postoperative hours. This scale consists of a 100-millimeter line, with 0 representing no symptoms and 100 representing the most severe symptoms ever experienced. Patients are asked to mark the intensity they feel on the line. A numerical value is then obtained by measuring the millimeter at which the mark appears.
Additional Analgesia | 24 hours
  The time when patients request painkiller for the first time despite their existing analgesia plan.
Nausea and Vomiting | 24 hours
  Nausea and vomiting according to Visual Analog Scale that can be observed at the 2nd and 24th postoperative hours.This scale consists of a 100-millimeter line, with 0 representing no symptoms and 100 representing the most severe symptoms ever experienced. Patients are asked to mark the intensity they feel on the line. A numerical value is then obtained by measuring the millimeter at which the mark appears.
Gas and Stool | 24 hours
  Time to pass gas or stool for the first time in the postoperative period.
Pittsburgh Sleep Quality Index score | 24 hours
  Evaluation of patients' sleep in the last month according to the Pittsburgh Sleep Quality Index score. The Pittsburgh Sleep Quality Index consists of seven components, each scored 0-3, yielding a global score of 0-21. Higher scores reflect poorer sleep quality, with a global score >5 indicating clinically significant sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Munire BABAYIGIT, Assoc. Prof., Study Director — Ankara Ataturk Sanatorium Research and Training Hospital
Locations (1):
- Ankara Ataturk Sanatorium Research and Training Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Kwon HM, Kim DH, Jeong SM, Choi KT, Park S, Kwon HJ, Lee JH. Does Erector Spinae Plane Block Have a Visceral Analgesic Effect?: A Randomized Controlled Trial. Sci Rep. 2020 May 21;10(1):8389. doi: 10.1038/s41598-020-65172-0. PMID 32439926
- [Background] Abu Elyazed MM, Mostafa SF, Abdelghany MS, Eid GM. Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Open Epigastric Hernia Repair: A Prospective Randomized Controlled Study. Anesth Analg. 2019 Jul;129(1):235-240. doi: 10.1213/ANE.0000000000004071. PMID 30801359
- [Background] Sorenstua M, Raeder J, Vamnes JS, Leonardsen AL. Evaluation of the Erector spinae plane block for postoperative analgesia in laparoscopic ventral hernia repair: a randomized placebo controlled trial. BMC Anesthesiol. 2024 May 29;24(1):192. doi: 10.1186/s12871-024-02566-x. PMID 38811911
- [Background] Elsharkawy H, Kolli S, Soliman LM, Seif J, Drake RL, Mariano ER, El-Boghdadly K. The External Oblique Intercostal Block: Anatomic Evaluation and Case Series. Pain Med. 2021 Nov 26;22(11):2436-2442. doi: 10.1093/pm/pnab296. PMID 34626112